CLINICAL TRIAL: NCT01605656
Title: A Mixed-Methods Approach to Understanding Factors Associated With Cervical Cancer Screening Utilization Among Low-Income, HIV-Positive Women
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2012-0240; R25T CA57730 (Registry Identifier: NCI)
Record Dates: First submitted 2012-05-18; First posted 2012-05-25 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Cancer Prevention; Cervix
Keywords: Cancer Prevention; Cervix; Questionnaires; Focus groups; Surveys; Interviews
MeSH Terms: interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Focus Groups + Interviews + Questionnaires: HIV-positive women recruited from the population of individuals seeking care at Thomas Street Health Center (TSHC) of the Harris County Hospital District (HCHD).
  Interventions: Behavioral: Cognitive Interview; Behavioral: Questionnaires; Behavioral: Focus Groups

INTERVENTIONS:
Behavioral: Cognitive Interview — A research staff member will use a questionnaire to ask about many different health and social topics. The cognitive interview should take up to 45 minutes to complete.
Behavioral: Questionnaires — Phase I: Completion of a questionnaire about age, education level, income, and general health behaviors. This questionnaire should take about 20 minutes to complete.
  Phase II: Completion of 2 questionnaires. The first questionnaire will ask about age, education level, income, and general health behaviors. This questionnaire should take about 20 minutes to complete.
  The second questionnaire will ask about many different health and social topics. This questionnaire should take up to 45 minutes to complete.
  Other Names: Surveys
Behavioral: Focus Groups — Phase I: There will be up to 8 women in each of the 5 focus groups.
  Participants asked questions about personal and clinic-related factors that might make it more difficult to receive pap smear screenings. Participants also asked to discuss what might make it easier or encourage women to receive pap smear screenings. The focus group discussion should last 60-90 minutes.

SUMMARY:
The goal of this study is to better understand the factors that might prevent HIV-positive women from having routine pap smear screenings. Researchers also want to learn what might make it easier or encourage women to have these screenings.

DETAILED DESCRIPTION:
Cognitive Interviews:

If you agree to take part in this study, you will be take part in a cognitive interview. A cognitive interview is a process that helps researchers test out questions on a few people so the questions can improved.

During the interview, a research staff member will use a questionnaire to ask you about many different health and social topics.

As the questions are read to you, please answer them, but also tell the research staff member what you're thinking. Please try to think out loud and say everything that comes to mind, whether it seems important or not. You will be asked how you came up with your answers and how you understood the questions. If any question seems unclear or hard to answer, please tell the research staff member. A member of the research staff will be taking notes during the interview.

The cognitive interview should take up to 45 minutes to complete.

Length of Study:

Your participation in this study will be over after you complete the cognitive interview.

This is an investigational study.

Up to 10 participants will be enrolled in this part of the study. All will take part at Thomas Street Health Center.

Phase I:

If you agree to take part in this study, you will complete a questionnaire about your age, education level, income, and general health behaviors. This questionnaire should take about 20 minutes to complete.

After completing the questionnaire, you will take part in a focus group discussion with other women who are patients at Thomas Street Health Center. There will be up to 8 women in each of the 5 groups.

In the focus group, you will be asked questions about personal and clinic-related factors that might make it more difficult to receive pap smear screenings. You will also be asked to discuss what might make it easier or encourage women to receive pap smear screenings. The focus group discussion should last 60-90 minutes.

The information discussed in the focus groups may be sensitive, so you will be asked to keep the information discussed in the group private.

Length of Study:

Your participation in this study will be over after you complete the questionnaire and participate in the focus group discussion.

This is an investigational study.

Up to 40 participants will be enrolled in this part of the study. All will take part at Thomas Street Health Center.

Phase II:

If you agree to take part in this study, you will complete 2 questionnaires. The first questionnaire will ask about your age, education level, income, and general health behaviors. This questionnaire should take about 20 minutes to complete.

The second questionnaire will ask about many different health and social topics. This questionnaire should take up to 45 minutes to complete.

Length of Study:

Your participation in this study will be over after you complete the 2 questionnaires.

This is an investigational study.

Up to 200 participants will be enrolled in this part of the study. All will take part at Thomas Street Health Center.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. Patient receiving HIV/AIDS care at Thomas Street Health Center
3. Female
4. 18 years of age or older
5. Able to provide written informed consent to participate

Exclusion Criteria:

1) Physically deemed ineligible based on medical (HIV related or other condition) or psychiatric condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-positive women seeking care at Thomas Street Health Center (TSHC) of the Harris County Hospital District (HCHD).
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
HIV Positive Women's Perceived Barriers to Cervical Cancer Screening | 1 day
  Participants rank Nominal Group Technique (NGT) items (cervical cancer screening barriers and strategies to improve screening) from 1-5 (1-least important: 5-most important). Once two coders have calculated rankings, the 5 items receiving the highest number of points will be deemed the 5 barriers to cervical cancer screening. Similarly, the 5 strategy-based items receiving highest number of points will be deemed essential strategies to improving cervical cancer screening at Thomas Street Health Center (TSHC).

CONTACTS AND LOCATIONS:
Overall Officials: Damon Vidrine, MS, DRPH, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Thomas Street Health Center, Harris County Hospital District, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org